CLINICAL TRIAL: NCT00929734
Title: Effect of ROsuvastatin Therapy on Peripheral Vasodilator Function, Inflammatory Markers and Pulmonary Function in Patients With StablE Chronic Obstructive Pulmonary Disease
Brief Title: Effect of Rosuvastatin Therapy in Patients With Stable Chronic Obstructive Pulmonary Disease
Acronym: RODEO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Akershus (Other)
Collaborators: AstraZeneca (Industry); Haukeland University Hospital (Other)
Responsible Party: Principal Investigator, Torbjorn Omland, Professor of Medicine, University Hospital, Akershus
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2009A2
Record Dates: First submitted 2009-06-26; First posted 2009-06-29 (Estimated); Results first posted 2015-10-08 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-09

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Inflammation; Atherosclerosis; Hydroxymethylglutaryl-coenzyme A Reductase Inhibitors
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Inflammation; Atherosclerosis | interventions — Rosuvastatin Calcium; Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rosuvastatin (Experimental)
  Interventions: Drug: Rosuvastatin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rosuvastatin — 10mg tablets, once daily in three months
  Other Names: Hydroxymethylglutaryl-CoA Reductase Inhibitor
  Arms: Rosuvastatin
Drug: Placebo — 1 tablet, once daily in three months
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate whether rosuvastatin improves measures of endothelial function, decreases measures of inflammation, and improves pulmonary function in patients with stable chronic obstructive pulmonary disease.

ELIGIBILITY:
Inclusion criteria:

* Stable COPD patients of both genders with no COPD exacerbations less than three weeks prior to inclusion
* COPD stage I to IV after the GOLD criteria (Global Initiative for Chronic Obstructive Lung Disease)
* Age between 40 and 80 years

Exclusion criteria:

* Diagnosed lung disease other than COPD, except chronic asthmatic bronchitis and mild bronchiectasis without or few physical signs (diagnosed by high resolution CT)
* History of or active coronary artery disease (CAD), cerebrovascular or peripheral vascular disease
* History of or clinically significant congestive heart failure, valvular heart disease, clinically significant arrhythmias or conduction delays
* History of uncontrolled arterial hypertension (defined as blood pressure above180/110 mmHg with or without the use of antihypertensive medication)
* Body mass index >40kg/m2
* History of diabetes mellitus, measured fasting glucose > 11 mmol/L
* History of Hypercholesterolemia, measured total cholesterol > 8 mmol/L
* Known poliomyelitis, motor neurone disease, cranial or temporal arteritis, stroke or myopathy
* Neutropenia, anemia (Hb < 8 g/100mL)
* History of chronic renal failure, serum creatinine > 176 micromol/L (2.0mg/dL)
* Creatine kinase > 3 times the upper limit of normal (ULN)
* Acute or chronic liver disease (serum transaminases > 3 times the ULN)
* Pregnancy (oral examination and blood test prior to inclusion)
* Active abuse of drugs or alcohol, poor compliance anticipated
* Statin use within the last 4 weeks prior to study start or previously clear indication for statin use
* Prior diagnosis of statin induced myopathy or hypersensitivity reaction to another hydroxymethylglutaryl-Coenzyme A-reductase inhibitor incl. Rosuvastatin
* History of malignant disease of any kind within 5 years prior to inclusion.
* History of uncontrolled hypothyroidism
* Participation in another pharmaceutical or medical device clinical trial study less than 4 weeks prior inclusion.
* Use concomitant of medications that are known to interact with Crestor. This includes the following medications: Warfarin and other coumarin (vitamin K antagonist) anticoagulants, Cyclosporin, Gemfibrozil and Antacid

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2010-03; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Torbjørn Omland, PhD, Principal Investigator — University Hospital, Akershus
Locations (1):
- Akershus University Hospital, Lørenskog, Akershus, Norway

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rosuvastatin | Placebo
Started | 49 | 50
Completed | 47 | 47
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Population: Complete case population
Groups:
- Rosuvastatin: Rosuvastatin 10mg tablet
- Placebo: Placebo tablet
- Total: Total of all reporting groups
Arm/Group | Rosuvastatin | Placebo | Total
Number analyzed (Participants) | 47 | 47 | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (5.5) | 63 (6.6) | 65 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 24 | 45
  Male | 26 | 23 | 49
BMI [Mean (Standard Deviation); unit: kg/m^2] | 23 (3.8) | 24 (4.1) | 24 (3.9)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 131 (17.7) | 135 (20.1) | 133 (18.9)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 79 (8.4) | 80 (10.3) | 80 (9.4)
Heart rate [Mean (Standard Deviation); unit: beats/min] | 68 (11.2) | 67 (10.9) | 67 (11.0)
History of hypertension [Number; unit: participants]
  Yes | 12 | 11 | 23
  No | 35 | 36 | 71
History of asthma [Number; unit: participants]
  Yes | 9 | 13 | 22
  No | 38 | 34 | 72
Pack-years [Mean (Standard Deviation); unit: pack-years] — Number of packs of cigarettes smoked per day by the number of years the person has smoked
  pack-years | 39 (16.1) | 35 (15.5) | 37 (15.8)
Current smoking [Number; unit: participants]
  Yes | 12 | 23 | 35
  No | 35 | 24 | 59
Haemoglobin [Mean (Standard Deviation); unit: g/dl] | 14.1 (1.4) | 14.0 (0.2) | 14.0 (1.2)
Estimated Glomerular Filtration Rate (eGFR) [Mean (Standard Deviation); unit: ml/min] — Renal function as calculated by the Cockcroft-Gault formula ((140- age) × bodyweight/serum creatinine) (× 0.85 for women))
  ml/min | 82.4 (19.6) | 90.1 (29.4) | 86.2 (25.1)
Leucocyte count [Mean (Standard Deviation); unit: cells*10^9/L] | 6.6 (1.4) | 6.9 (1.7) | 6.7 (1.6)
High-sensitivity C-reactive protein [Median (Inter-Quartile Range); unit: mg/L] — Acute-phase reactant used in cardiovascular risk assessment
  mg/L | 1.4 [0.8 to 3.7] | 1.8 [1.0 to 4.4] | 1.7 [0.8 to 3.8]
Interleukin 6 [Median (Inter-Quartile Range); unit: pg/mL] | 4.1 [2.9 to 5.3] | 3.4 [2.7 to 4.7] | 3.7 [2.7 to 5.1]
Glucose [Mean (Standard Deviation); unit: mmol/L] | 5.0 (0.6) | 5.1 (0.7) | 5.0 (0.6)
Cholesterol [Mean (Standard Deviation); unit: mmol/L] | 5.5 (0.9) | 5.7 (1.1) | 5.6 (1.0)
LDL-C [Mean (Standard Deviation); unit: mmol/L] | 3.3 (0.8) | 3.5 (0.9) | 3.4 (0.9)
HDL-C [Mean (Standard Deviation); unit: mmol/L] | 1.8 (0.1) | 1.8 (0.1) | 1.8 (0.5)
Triglycerides [Mean (Standard Deviation); unit: mmol/L] | 1.0 (0.4) | 1.1 (0.5) | 1.1 (0.4)
Forced expiratory volume at one second (FEV1) [Mean (Standard Deviation); unit: Liter] | 1.4 (0.6) | 1.5 (0.7) | 1.4 (0.6)
FEV1, % of predicted [Mean (Standard Deviation); unit: Percent predicted value] | 48.3 (18.9) | 52.1 (18.8) | 50.2 (18.9)
FEV1/FVC [Mean (Standard Deviation); unit: Percent of FVC] — Forced vital capacity (FVC)
  Percent of FVC | 47 (13.8) | 49 (11.8) | 48 (12.8)
Antihypertensive treatment [Number; unit: participants]
  Yes | 12 | 10 | 22
  No | 35 | 37 | 72
Inhaled corticosteroids [Number; unit: participants] — including long acting beta agonists (LABA)
  participants
    Yes | 36 | 34 | 70
    No | 11 | 13 | 24
Long acting beta agonists [Number; unit: participants]
  Yes | 2 | 3 | 5
  No | 45 | 44 | 89
Long acting muscarinic antagonists [Number; unit: participants]
  Yes | 30 | 27 | 57
  No | 17 | 20 | 37
Anti-inflammatory treatment [Number; unit: participants]
  Yes | 2 | 0 | 2
  No | 45 | 47 | 92
Oestrogen treatment [Number; unit: participants]
  Yes | 4 | 3 | 7
  No | 43 | 44 | 87

OUTCOME MEASURES:

1. Primary Outcome: Relative Change in Reactive Hyperemia Index (RHI)
Description: Endothelial function assessed with peripheral arterial tonometry, expressed as the reactive hyperemia index (RHI) as a marker for subclinical atherosclerosis and future cardiovascular risk assessment.
Time Frame: Baseline to 3 months
Population: Complete case analysis
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Rosuvastatin | Placebo
Number analyzed (Participants) | 47 | 47
percent change | 6.65 [1.80 to 15.11] | -1.27 [-8.33 to 5.79]
Statistical Analysis 1: Comparison: Rosuvastatin vs Placebo; Test type: Superiority or Other; p = 0.292, ANCOVA

2. Secondary Outcome: Relative Change in FEV1
Time Frame: Baseline to 3 months
Population: Complete case analysis
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Rosuvastatin | Placebo
Number analyzed (Participants) | 47 | 47
percent change | 2.6 [-2.2 to 7.5] | -1.1 [-4.7 to 2.5]
Statistical Analysis 1: Comparison: Rosuvastatin vs Placebo; Test type: Superiority or Other; p = 0.462, ANCOVA

3. Secondary Outcome: Relative Change in High-sensitivity C-reactive Protein
Time Frame: Baseline to 3 months
Population: Complete case analysis
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Rosuvastatin | Placebo
Number analyzed (Participants) | 47 | 47
percent change | -20.0 [-45.8 to 14.3] | 11.0 [-35.1 to 93.3]
Statistical Analysis 1: Comparison: Rosuvastatin vs Placebo; Test type: Superiority or Other; p = 0.017, ANCOVA — ANCOVA with natural logarithm of hs-CRP (ln hs-CRP)

4. Secondary Outcome: Relative Change in Interleukin 6
Time Frame: Baseline to 3 months
Population: Complete case analysis
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Rosuvastatin | Placebo
Number analyzed (Participants) | 47 | 47
percent change | 8 [-20 to 43.8] | 30 [0 to 52.2]
Statistical Analysis 1: Comparison: Rosuvastatin vs Placebo; Test type: Superiority or Other; p = 0.028, ANCOVA — ANCOVA with natural logarithm of interleukin 6 (ln IL6)

ADVERSE EVENTS:
Time Frame: 3 months
Description: Data are presented for all patients with adverse event registration (patient diary).
  The 2 patients lost to follow-up in the rosuvastatin arm had missing adverse event data.
  2 of 3 patients without control investigation in the placebo arm withdrew, but provided adverse event data.
Arm/Group | Rosuvastatin | Placebo
Serious Adverse Events (participants affected / at risk) | 4/47 | 3/49
Other Adverse Events (participants affected / at risk) | 12/47 | 21/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rosuvastatin (N=47) | Placebo (N=49)
Acute exacerbation of chronic obstructive pulmonary disease (AECOPD) (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) — Hospitalization for AECOPD
Hypophysis apoplexia (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rosuvastatin (N=47) | Placebo (N=49)
AECOPD (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 12 (12)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Nervous system disorders) | 2 (2) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Orthostatic vertigo (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Ankle edema (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Vascular disorders) | 0 (0) | 1 (1)
Urinary retension (Renal and urinary disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Cold (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No